CLINICAL TRIAL: NCT01145885
Title: Investigation of the Metabolism, Excretion and Pharmacokinetics of an Openlabel Single Dose of 300 mg [14C]Volasertib Administered Intravenously in Patients With Various Solid Tumours With a Possible Extension Phase With Nonlabelled Drug
Brief Title: BI 6727 (Volasertib) Human ADME Trial in Various Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.23; 2009-018199-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727

ARMS (1):
- BI 6727 (Experimental): BI 6727 cycles in every 21 days
  Interventions: Drug: BI 6727

INTERVENTIONS:
Drug: BI 6727 — PLK-1 inhibitor

SUMMARY:
Investigation of absorption, distribution, metabolism and excretion (ADME) and assessment of safety, tolerability and preliminary therapeutic effects of [14C]volasertib in patients with advanced solid tumours.

ELIGIBILITY:
Inclusion criteria:

* Inclusion Criteria 1. Patients with histologically or cytologically confirmed diagnosis of advanced, non resectable and / or metastatic solid tumour
* Inclusion Criteria 2. Male
* Inclusion Criteria 3. Age >=18 and =<70 years
* Inclusion Criteria 4. Written informed consent
* Inclusion Criteria 5. Eastern Cooperative Oncology Group (ECOG) performance score =<2
* Inclusion Criteria 6. Recovery from Common Terminology Criteria for Adverse Events (CTCAE) Grade >=2 therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapy

Exclusion criteria:

* Exclusion Criteria 1. Serious concomitant non-oncological disease considered by the investigator
* Exclusion Criteria 2. Active infectious disease
* Exclusion Criteria 3. Viral hepatitis, Human Immunodeficiency Virus (HIV) infection
* Exclusion Criteria 4. Clinical evidence of active brain metastasis during the past 6 months
* Exclusion Criteria 5. Second malignancy currently requiring active therapy
* Exclusion Criteria 6. Absolute neutrophil count less than 1,500/mm3
* Exclusion Criteria 7. Platelet count less than 100,000/mm3
* Exclusion Criteria 8. Total bilirubin greater than 1.5 mg/dL
* Exclusion Criteria 9. Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Exclusion Criteria 10. Serum creatinine greater than 1.5x Upper Limit of Normal (ULN).
* Exclusion Criteria 11. Known history of QT/QTcF-prolongation
* Exclusion Criteria 12. Patients who are sexually active and having a partner with childbearing potential and unwilling to use a medically acceptable method of contraception
* Exclusion Criteria 13. Treatment with other investigational drugs or participation in another clinical trial
* Exclusion Criteria 14. Chemo-, radio- immuno-, or molecular-targeted cancer-therapy within the past four weeks prior to start of therapy or concomitantly with this trial. This restriction does not apply to steroids and bisphosphonates.
* Exclusion Criteria 15. Alcohol abuse
* Exclusion Criteria 16. Life expectancy less than 12 weeks
* Exclusion Criteria 17. Potent Cytochrome P450 enzyme (CYP) 3A4 and P-glycoprotein inhibitors or inducers
* Exclusion Criteria 18. History of allergy/hypersensitivity

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1230.23.36001 Boehringer Ingelheim Investigational Site, Budapest, Hungary

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants entered the first treatment cycle, if they experienced clinical benefit from the first treatment course they could continue into further treatment courses.
Groups:
- Volasertib: Participants received 300mg 14C volasertib ((14C) BI 6727) as a single dose via intravenous infusion on day 1 of the the first treatment cycle (21 days).
Period: Overall Study
Arm/Group | Volasertib
Started | 7
Completed | 0
Not Completed | 7
Not completed — Progressive Disease | 7

BASELINE CHARACTERISTICS:
Population: Treated set which included all patients who were dispensed study medication and were documented as having taken at least 1 dose of investigational treatment.
Arm/Group | Volasertib
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Individual Time Course Profiles of 14C-radioactivity in Whole Blood and Plasma: Cmax of 14C Labelled Volasertib
Description: Individual time course profiles of 14C-radioactivity in whole blood and plasma: Cmax of 14C labelled Volasertib.
Time Frame: Whole blood: Pre-dose (-0.5 hours (h)) and 1.0h, 1.983h, 4h, 6h, 8h and 24h after start of the 2h drug infusion.Plasma: Pre-dose (-0.5h) and 1.0h, 1.983h, 4h, 6h, 8h, 24h,48h. 96h, 168h and 336h after start of drug infusion.
Population: Pharmacokinetic (PK) set which included all evaluable patients in the treated set who provided at least 1 observation for at least 1 primary PK endpoint and did not undergo important protocol violations relevant to the evaluation of PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Volasertib 14C 300 mg: Participants received 300mg 14C volasertib ((14C) BI 6727) as a single dose via intravenous infusion on day 1 of the the first treatment cycle (21 days).
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol/L
  Whole Blood | 1746 (18.0)
  Plasma | 1150 (14.7)

2. Primary Outcome: Individual Time Course Profiles of 14C-radioactivity in Urine: Cumulative Fraction of 14C-ratioactivity Excreted in Urine
Description: Percentage of administered dose excreted in urine as 14C-radioactivity over time
Time Frame: Every 24 hours, up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
Percentage of dose
  0-24 hours | 4.21 (33.8)
  0-168 hours | 11.7 (23.9)
  0-336 hours | 15.6 (22.5)
  0-504 hours | 18.1 (21.9)

3. Primary Outcome: Individual Time Course Profiles of 14C-radioactivity in Faeces: Cumulative Fraction of 14C-radioactivity Excreted in Faeces
Description: Percentage of administered dose excreted in faeces as 14C-radioactivity over time
Time Frame: Every 24 hours, up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
Percentage of dose
  0-24 hours | 0.680 (433)
  0-168 hours | 24.4 (46.2)
  0-336 hours | 36.7 (33.0)
  0-504 hours | 42.5 (29.3)

4. Primary Outcome: Individual Time Course Profiles of Volasertib and CD 10899 in Plasma: Cmax of Volasertib and CD 10899 (a Metabolite of Volasertib).
Description: Individual time course profiles of volasertib (BI 6727) and a metabolite of volasertib (CD 10899), in plasma: Cmax of Volasertib and CD 10899.
Time Frame: Plasma: Pre-dose (-0.5h) and 1.0h, 1.983h, 4h, 6h, 8h, 24h,48h. 96h, 168h and 336h after start of drug infusion.
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol/L
  Volasertib (1.983 hours) | 926 (17.8)
  CD 10899 (6 hours) | 9.92 (29.8)

5. Primary Outcome: Individual Time Course Profile of Volasertib in Urine:Cumulative Fraction of Volasertib Excreted in Urine
Description: Percentage of administered dose excreted in urine as volasertib (BI 6727) over time
Time Frame: Every 24 hours, up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
Percentage of dose
  0-24 hours | 3.24 (31.6)
  0-168 hours | 7.57 (28.4)
  0-336 hours | 9.14 (28.7)
  0-504 hours | 9.89 (29.2)

6. Primary Outcome: Individual Time Course Profile of CD 10899 in Urine: Cumulative Amount of CD 10899 Excreted in Urine
Description: Cumulative amounts of CD 10899, a metabolite of volasertib, excreted in urine over time
Time Frame: Every 24 hours, up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol
  0-24 hours | 1240 (54.9)
  0-168 hours | 5670 (37.3)
  0-336 hours | 7580 (34.4)
  0-504 hours | 8490 (33.6)

7. Primary Outcome: Rate and Extent of Excretion Mass Balance Based on the Total Radioactivity in Urine and Faeces: Cumulative Fraction of Excretion 504 Hours After Start of Drug Infusion.
Description: Cumulative Percentage of 14C-radioactivity excreted in urine and faeces at 504 hours after start of drug infusion related to total [14C] volasertib administered.
Time Frame: up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
Percentage of dose
  Urine | 18.1 (21.9)
  Faeces | 42.5 (29.3)

8. Primary Outcome: Cmax of Volasertib and CD 10899 in Plasma
Description: Maximum measured concentration of volasertib and CD 10899, a metabolite of volasertib, in plasma (Cmax).
Time Frame: 30 minutes (min) before start of infusion and 1 hour (h), 1h 59min, 4h, 6h, 8h, 24h, 48h, 96h, 168h and 336h after start of infusion
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol/L
  Volasertib | 926 (17.8)
  CD 10899 | 11.1 (24.5)

9. Primary Outcome: AUC0-inf of Volasertib and CD10899 in Plasma
Description: Area under the concentration-time curve of volasertib and CD 10899, a metabolite of volasertib, in plasma over the time interval from 0 to infinity (AUC0-inf).
Time Frame: as for outcome 8
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol*h/L
  Volasertib | 11400 (22.3)
  CD 10899 | 1500 (16.8)

10. Primary Outcome: CL/R of Volasertib and CD 10899 in Urine
Description: Renal clearance of the analyte in urine (CL/R) within the time interval 0 hours to 504 hours of volasertib and CD 10899, a metabolite of volasertib.
Time Frame: Every 24 hours, up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
mL/min
  Volasertib | 68.5 (23.2)
  CD 10899 | 102 (26.8)

11. Primary Outcome: Ae(0-tz) of Volasertib and CD 10899 in Urine
Description: Amount of analyte eliminated in urine within the time interval 0 hours to last quantifiable data point (Ae(0-tz)) for volasertib and CD 10899, a metabolite of volasertib.
Time Frame: Every 24 hours, up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol
  Volasertib | 45800 (29.3)
  CD 10899 | 8490 (33.6)

12. Primary Outcome: AUC0-tz of 14C Radioactivity in Plasma and Whole Blood
Description: Area under the concentration-time curve of 14C radioactivity in plasma and whole blood over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: 30 minutes (min) before start of infusion and 1 hour (h), 1h 59min, 4h, 6h, 8h, 24h, 48h, 96h, 168h and 336h after start of infusion for plasma; 30 min before start of infusion and 1h, 1h 59min, 4h, 6h, 8h and 24h after start of infusion for whole blood
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol*h/L
  Plasma | 4450 (57.6)
  Whole blood | 8810 (26.5)

13. Primary Outcome: Ae(0-tz) of 14C Radioactivity in Urine
Description: Amount of analyte eliminated in urine within the time interval 0 to to the last quantifiable data point (Ae(0-tz)) of 14C radioactivity
Time Frame: Every 24 hours, up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol | 84000 (22.1)

14. Primary Outcome: Ae,Faeces(0-tz) of 14C Radioactivity
Description: Amount of analyte excreted in faeces within the time interval 0 to to the last quantifiable data point (Ae(0-tz)) of 14C radioactivity
Time Frame: Every 24 hours, up to 504 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
nmol | 197000 (29.1)

15. Primary Outcome: Time Dependency of Cblood Cells/Cplasma Ratio and Cblood/Cplasma Ratio of 14C-radioactivity
Description: Time dependency of Cblood cells/Cplasma ratio and Cblood/Cplasma ratio of 14C-radioactivity.
Time Frame: 1.983 hours and 6 hours
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 6
Ratio
  Cblood/Cplasma ratio: 1.983 hours | 1.52 (9.67)
  Cblood/Cplasma ratio: 6 hours | 1.54 (9.30)
  Cblood cells/Cplasma ratio: 1.983 hours | 2.66 (13.8)
  Cblood cells/Cplasma ratio: 6 hours | 2.76 (18.8)

16. Primary Outcome: Elucidation of Metabolite Structures and Identification of Major Metabolites in Plasma, Urine, and Faeces
Description: Elucidation of mb structures and identification of major metabolites in plasma, urine, and faeces. This endpoint was not analysed in the study report.
  The contribution of volasertib and the metabolite CD 10899 to total radioactivity in plasma in the time interval 0 to 8 h after drug administration supports the suggestion that other metabolites in addition to CD 10899 are present in plasma. However, different methods used for the quantification of volasertib and CD 10899 (HPLC MS/MS) and total 14C-radioactivity (liquid scintillation counting) have to be taken into account for the interpretation of the difference between total 14C-radioactivity and analysis of volasertib and CD 10899 in plasma and the plasma metabolite pattern remains to be categorized.
Time Frame: 3 weeks
Population: This endpoint was not analyzed. Please refer to the description for the explanation.
Arm/Group | Volasertib 14C 300 mg
Number analyzed (Participants) | 0

17. Secondary Outcome: Percentage of Participants With Drug Related Adverse Events
Description: Percentage of participants with drug related adverse events (AEs)
Time Frame: From first intake of study drug until 21 days after last intake of the study drug, up to 63 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Groups:
- Volasertib 300mg: Participants received 300mg non-radiolabelled volasertib (BI 6727) via intravenous infusion on day 1 of each 21-day treatment cycle, in treatment cycles 2 or 3.
- Volasertib 250mg: Participants received 250mg non-radiolabelled volasertib (BI 6727) via intravenous infusion on day 1 of each 21-day treatment cycle, in treatment cycles 2 or 3.
Arm/Group | Volasertib 14C 300 mg | Volasertib 300mg | Volasertib 250mg
Number analyzed (Participants) | 7 | 3 | 2
Percentage of participants | 100.0 | 100.0 | 100.0

18. Secondary Outcome: Percentage of Participants With Clinically Relevant Abnormalities for Clinical Assessments, ECG, Vital Signs and Laboratory Tests
Description: Percentage of participants with clinically relevant abnormalities for clinical assessments, electrocardiogram (ECG), vital signs and clinical laboratory test parameters. New abnormal findings or worsening of baseline conditions were reported as adverse events.
Time Frame: From first intake of study drug until 21 days after last intake of the study drug, up to 63 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Volasertib 14C 300 mg | Volasertib 300mg | Volasertib 250mg
Number analyzed (Participants) | 7 | 3 | 2
Percentage of participants | 0.0 | 0.0 | 0.0

19. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: The endpoint tumour response was was analysed as the percentage of participants with clinical benefit after each treatment cycle based on the Investigator's response assessment (with clinical assessment being conducted after every cycle and radiological assessment at the Investigator's discretion).
Time Frame: 21, 42 and 63 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Volasertib 14C 300 mg | Volasertib 300mg | Volasertib 250mg
Number analyzed (Participants) | 7 | 3 | 2
Percentage of participants
  End of cycle 1 (21 days): Clinical Benefit=No | 42.9 | 0.0 | 0.0
  End of cycle 1 (21 days): Clinical Benefit=Yes | 57.1 | 0.0 | 0.0
  End of cycle 2 (42 days): Clinical Benefit=No | 0.0 | 66.7 | 100.0
  End of cycle 2 (42 days): Clinical Benefit=Yes | 0.0 | 33.3 | 0.0
  End of cycle 3 (63 days): Clinical Benefit=No | 0.0 | 0.0 | 100.0
  End of cycle 3 (63 days): Clinical Benefit=Yes | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first intake of study drug until 21 days after last intake of the study drug, up to 63 days
Groups:
- Volasertib 14C 300mg; Volasertib: Participants received 300mg 14C volasertib ((14C) BI 6727) as a single dose via intravenous infusion on day 1 of the the first treatment cycle (21 days).
- Total_Volasertib 300: Participants received 300mg 14C volasertib ((14C) BI 6727) as a single dose via intravenous infusion on day 1 of the the first treatment cycle (21 days) and patient who continued into further treatment cycles and received 300mg non-radiolabelled volasertib (BI 6727) via intravenous infusion on day 1 of each 21-day treatment cycle.
- Volasertib 250mg: Participants received 300mg non-radiolabelled volasertib (BI 6727) via intravenous infusion on day 1 of each 21-day treatment cycle, in treatment cycles 2 or 3.
Arm/Group | Volasertib 14C 300mg | Volasertib 300mg | Total_Volasertib 300 | Volasertib 250mg | Volasertib
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/3 | 1/7 | 0/2 | 1/7
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 7/7 | 2/2 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 14C 300mg (N=7) | Volasertib 300mg (N=3) | Total_Volasertib 300 (N=7) | Volasertib 250mg (N=2) | Volasertib (N=7)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 14C 300mg (N=7) | Volasertib 300mg (N=3) | Total_Volasertib 300 (N=7) | Volasertib 250mg (N=2) | Volasertib (N=7)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 5 | 1 | 5
Leukopenia (Blood and lymphatic system disorders) | 5 | 3 | 6 | 2 | 6
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 4 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 3 | 6 | 2 | 6
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to improper mixing of the infusion solution, the actual dose administered could not reliably be determined for one patient so the PK data for this patient were excluded from the analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.